CLINICAL TRIAL: NCT04779658
Title: Essure Removal for Device-attributed Symptoms: Quality of Life Evaluation Before and After Surgical Removal
Brief Title: Laparoscopic Essure Device Removal
Acronym: ESSURE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0087
Record Dates: First submitted 2021-02-18; First posted 2021-03-03 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-02

CONDITIONS: Contraception
Keywords: Essure device removal; Quality of life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In recent years, several symptoms have been attributed to Essure, including pelvic pain and other general symptoms. Consequently, an increasing number of patients request Essure removal for alleged adverse reactions to the device.

Study Objective: To evaluate the quality of life of patients who underwent Essure_ device removal and morbidity of this surgery.

Design: Prospective observational cohort study. Setting: Academic hospitals of La Conception, Marseille, and Arnaud-de-Villeneuve, Montpellier, France.

Patients: Women who underwent Essure_ device removal by salpingectomy, between February 2017 and August 2018.

Methods : The following information have been collected during preoperative clinics: demographic data, medical history, clinical symptoms attributed to the Essure device, time between Essure sterilization and early symptoms, time between the beginning of symptoms and surgical removal. Follow-up visits have benne scheduled at one month and three months post-operation. The evolution of symptoms was collected during the follow-up visit at three months based on clinical reports and a dedicated questionnaire. Evaluation of Quality of life have been evaluated thanks to SF36 and HAD questionnaires. Alle these patients will be contacted by phone call to assess to evolution of symptoms and to complete SF 36 and HAD questionnaires.

Hypothesis : Recovery of symptoms due to ESSURE device and improvement of quality of life after surgery.

ELIGIBILITY:
Inclusion criteria:

* age >18 years old
* symptoms related to ESSURE device
* salpingectomy for ESSURE removal

Exclusion criteria:

- Exclusion criteria were failure to perform a complete removal of the Essure and second surgery to remove fragments left behind from a previous procedure.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women who underwent Essure_ device removal by salpingectomy, between February 2017 and August 2018.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-29 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of quality of life after ESSURE removal | Preoperative
  Evaluation of quality of life after ESSURE removal by SF 36 questionnaire Preoperative questionnaires will be collected from medical record. Patients will be contacted by phone call to answer to this questionnaire for the long term follow-up
Evaluation of quality of life after ESSURE removal | three-months post-operative
  Evaluation of quality of life after ESSURE removal by SF 36 questionnaire three-months post-operative questionnaires will be collected from medical record. Patients will be contacted by phone call to answer to this questionnaire for the long term follow-up

SECONDARY OUTCOMES:
Evaluation of morbidity of ESSURE removal | 1 day
  description of per et postoperative complications (patient's medical record and by phone call)

CONTACTS AND LOCATIONS:
Overall Officials: Martha DURAES, Md, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC